CLINICAL TRIAL: NCT03236415
Title: Comparative Response to Vascular Injury in Patients With Diabetes Mellitus: An OCT Study of BVS Versus Xience DES
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Global sales of the Absorb BVS halted effective September 14, 2017.
Sponsor: Ottawa Heart Institute Research Corporation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20170128-01H
Record Dates: First submitted 2017-06-19; First posted 2017-08-01 (Actual); Last update posted 2017-10-19 (Actual); Status verified 2017-08

CONDITIONS: Coronary Artery Disease; Diabetes Mellitus
MeSH Terms: conditions — Coronary Artery Disease; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Xience Drug Eluting Stent (Active Comparator): Patients with diabetes mellitus will be randomized to receive either a Xience drug eluting stent or an ABSORB bioresorbable vascular scaffold for treatment of obstructive coronary artery disease
  Interventions: Device: Xience Drug Eluting Stent
- ABSORB Bioresorbable Vascular Scaffold (Active Comparator): Patients with diabetes mellitus will be randomized to receive either a Xience drug eluting stent or an ABSORB bioresorbable vascular scaffold for treatment of obstructive coronary artery diseasee
  Interventions: Device: ABSORB Bioresorbable Vascular Scaffold

INTERVENTIONS:
Device: Xience Drug Eluting Stent — Patients will undergo insertion of a drug eluting stent with assessment of strut coverage using optical coherence tomography at 4 to 6 weeks after implantation.
  Arms: Xience Drug Eluting Stent
Device: ABSORB Bioresorbable Vascular Scaffold — Patients will undergo insertion of a bioresorbable vascular scaffold with assessment of strut coverage using optical coherence tomography at 4 to 6 weeks after implantation.
  Arms: ABSORB Bioresorbable Vascular Scaffold

SUMMARY:
Stents are used at centers around the world to unblock the arteries of the heart. These stents are usually made of metal and remain permanently within the blood vessel wall. Newer developments in the stent technology has led to stent scaffolds that can be reabsorbed over time. Patients with diabetes are prone to more complex blockages in the heart arteries which can be more difficult to treat. The purpose of this study is to compare the difference of how arteries heal early when metal stents or resorbable stents are used in patients with diabetes.

DETAILED DESCRIPTION:
Coronary revascularization by percutaneous coronary intervention (PCI) is the dominant strategy in patients with obstructive coronary artery disease (CAD). Traditionally, PCI is performed with implantation of one or more permanent metallic stents which act as a scaffold for arterial recoil and, in the case of drug eluting stents (DES), provide a platform for delivery of anti-proliferative agents. A recent innovation in coronary stent technology is the advent of a bioresorbable vascular scaffold (BVS) - a poly L-lactide (PLLA) scaffold covered with a poly D,L-lactide coating which elutes everolimus. Bioresorption occurs by de-esterification of the long chains of PLLA into small particles which are then phagocytosed by macrophages. Within two years, the BVS is completely resorbed and vasomotor reactivity of the blood vessel is restored.

Patients with diabetes mellitus (DM) represent a clinically challenging population - having an increased incidence of complex CAD as well as higher rates of stent thrombosis (ST) and in-stent restenosis (ISR) following PCI. ST occurs most frequently in the first thirty days following stent implantation and is prevented by effective antiplatelet medications, optimization of stent deployment and by rapid reendothelialization (RE) of the device. Notably, patients with DM have delayed RE following stent implantation which results in a marked increase in risk of ST. Thus, patients with DM in particular are in need of devices that result in rapid establishment of stent coverage by optimizing the response to vascular injury.

Our study aims to answer the question: "Are there important differences in early healing between BVS and DES in patients with DM?" Our study hypothesis is that a BVS platform will enhance vascular healing resulting in greater strut coverage by 6 weeks in patients with DM.

This is a single centre, interventional, prospective cohort study which will be conducted between July 2017 and July 2019. A total of 52 patients will be recruited for participation in this study. Stable patients with diabetes will undergo randomization to either BVS or DES in the first target lesion using optical coherence tomography (OCT) at the time of the index procedure. Subsequently, patients will undergo staged PCI at four or six weeks (sub-randomization) of the second lesion with OCT evaluation of the initially implanted device to determine the percent of uncovered struts.

ELIGIBILITY:
Inclusion Criteria:

1. Stable patients with diabetes mellitus
2. Two or more stenoses in a major epicardial native coronary artery
3. An indication for PCI (i.e. >70% on angiography or fractional flow reserve (FFR) <0.8)
4. Coronary anatomy suitable for a BVS

Exclusion Criteria:

1. Unwillingness or inability to provide informed consent.
2. ST-elevation myocardial infarction
3. Hemodynamic instability

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-08 (Estimated); Primary Completion 2019-07 (Estimated); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
Percentage of uncovered struts at time of follow-up optical coherence tomography | 4 to 6 weeks
  The primary outcome will be the percent of uncovered struts analyzed at 5mm segments using a standardized protocol for optical coherence tomography at time of staged percutaneous coronary intervention procedure

SECONDARY OUTCOMES:
Late lumen loss | 4 to 6 weeks
  Assessment of standardized lumen area at 5mm increments
Neointimal area:artery area | 4 to 6 weeks
  Assessment of standardized neointimal area:artery area at 5mm increments
Strut malapposition | 4 to 6 weeks
  Assessment of strut malapposition as a percentage of total struts
In-stent restenosis | 4 to 6 weeks
  Binary in-stent restenosis defined as greater than 50% in-stent lumen loss
Target lesion revascularization | 4 to 6 weeks
  Any intervention within 5mm of the study device
Major adverse cardiac events | 4 to 6 weeks
  A composite of death, myocardial infarction or stroke

OTHER OUTCOMES:
Subgroup analysis between 4 and 6 weeks | 4 to 6 weeks
  A subgroup analysis between four and six weeks will be performed to study the gradation of intimal response during early vascular healing

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Hibbert, MD PhD, Principal Investigator — Ottawa Heart Institute Research Corporation

IPD SHARING:
Plan to Share IPD: No